CLINICAL TRIAL: NCT00620217
Title: Therapeutic Angiogenesis Using Human VEGF-A165/bFGF Plasmid Injected Percutaneously Into the Ischemic Myocardium of "No-option" Coronary Artery Disease Patients; Double-blind Placebo Controlled Study
Brief Title: Angiogenesis Using VEGF-A165/bFGF Plasmid Delivered Percutaneously in No-option CAD Patients; a Controlled Trial
Acronym: VIF-CAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Center of Oncology, Warsaw, Poland (Unknown); Medical University of Warsaw (Other); Ministry of Scientific Research and Information Technology, Poland (Other Government); Polpharma Foundation for Development of Polish Pharmacy and Medicine (Unknown)
Responsible Party: Prof. Witold Ruzyllo, Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBZ-KBN-099/P05/01
Record Dates: First submitted 2008-02-04; First posted 2008-02-21 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Coronary Artery Disease
Keywords: heart ischemia; coronary artery disease; plasmid; VEGF; FGF; percutaneous; gene therapy; SPECT; nuclear magnetic resonance
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): intramyocardial injection of bicistronic VEGF-A165/bFGF plasmid
  Interventions: Genetic: intramyocardial injection of VEGF-A165/bFGF:placebo plasmid
- 2 (Placebo Comparator): intramyocardial injection of placebo plasmid
  Interventions: Genetic: intramyocardial injection of VEGF-A165/bFGF:placebo plasmid

INTERVENTIONS:
Genetic: intramyocardial injection of VEGF-A165/bFGF:placebo plasmid — The plasmid will be given at a total dose of 0.5 mg, 10 injections of 0,2 ml each into the region of reversible ischemia. The process of injecting the solution into each of ten points within the ischemic zone will take 20 to 40 seconds to minimize muscle disruption

SUMMARY:
Achieving therapeutic angiogenesis with gene therapy using a plasmid coding human VEGF-A165/bFGF injected into ischemic myocardium of refractory coronary artery disease patients, employing a percutaneous catheter-based technique- a double-blind placebo controlled study.

Some patients with persistent coronary artery disease cannot be effectively treated using methods available today ("no-option" patients). It is currently evident that an emerging therapy for them might be the stimulation of neoangiogenesis in the area of ischemic myocardium using growth factor genes. Agents attracting greatest interest are FGF (fibroblast growth factor) and VEGF (vascular-endothelial growth factor). A number of methods have been tested to deliver these agents to the area of interest.

Basic research has revealed that potent forms of angiogenic growth factors are the basic FGF (bFGF) and VEGF type A. Most clinical research on therapeutic angiogenesis is done using one of these two growth factors. This is to our knowledge the first clinical study using bicistronic VEGF-A 165/bFGF plasmid.

Patient population will comprise CCS III and CCS IV coronary artery disease patients who cannot be treated with standard revascularization methods. In the course of study we shall attempt to analyze the efficacy of therapeutic plasmid-induced angiogenesis in terms of myocardial perfusion increase and clinical symptom improvement. The feasibility and safety of plasmid delivery method will also be assessed. A percutaneous catheter-based technique (Myo-Star, Johnson & Johnson®) is used for plasmid delivery.

All patients enrolled will receive optimal medical treatment as judged by treating physician. An effort will be made to modify medical therapy during the study course only for clear reasons.

Standard angiography and ventriculography will be performed prior to plasmid injection therapy. Ischemic area of interest will be identified on inclusion by SPECT. Cardiac nuclear magnetic resonance (cNMR) with adenosine will also be performed to assess heart morphology, function and perfusion. Next, injections will be performed according to protocol.

Follow-up visits will be performed at month 4 and month 12 after injection therapy.

A change in myocardial perfusion at rest and on dipyridamole-stress SPECT evaluation after injection therapy will be the primary measure of efficacy. Changes in exercise tolerance will also be monitored along with a number of other efficacy and safety parameters.

DETAILED DESCRIPTION:
Aim of the Study:

Achieving therapeutic angiogenesis with gene therapy using a plasmid coding human VEGF-A165/bFGF injected into ischemic myocardium of refractory coronary artery disease patients, employing a percutaneous catheter-based technique- a double-blind placebo controlled study.

A large group of patients with severe persistent symptoms of coronary artery disease cannot be effectively treated using the methods available today - they are sometimes described as "no-option" patients. It is currently evident that a promising emerging therapy for these patients might be the stimulation of neoangiogenesis in the area of ischemic myocardium, which generally requires the use of growth factors. Different methods and different growth factors have been used in experiments testing this approach. The two agents attracting the greatest interest of researchers are naturally FGF (fibroblast growth factor) and VEGF (vascular-endothelial growth factor). A number of methods, both in animal and human experiments, have also been tried to deliver these agents effectively to the area of interest and to ensure their prolonged action in target tissue.

Basic research has revealed that the most potent forms of angiogenic growth factors are the basic FGF (bFGF) and VEGF type A, especially in its 165 amino-acid form (VEGF-A 165) For this reason most clinical research on therapeutic angiogenesis is done using one of these two growth factors. This is to our knowledge the first clinical study using bicistronic VEGF-A 165/bFGF plasmid.

Study design:

The aim of the study is to achieve therapeutic angiogenesis with gene therapy using a bicistronic plasmid encoding human VEGF-A165/bFGF (pVIF) injected into ischemic myocardium. A percutaneous catheter-based technique (Myo-Star, Johnson & Johnson®) is used for plasmid delivery. The study is planned as a double-blind prospective placebo controlled trial.

The patient population will comprise of CCS III and CCS IV coronary artery disease patients who cannot be treated with any standard revascularization methods ("no-option" patients). In the course of the study we shall attempt to analyze the efficacy of therapeutic plasmid-induced angiogenesis in terms of myocardial perfusion increase and clinical symptom improvement. The feasibility and safety of plasmid delivery method will also be assessed.

The study will be conducted in accordance with the Declaration of Helsinki, 1964, with later amendments.

Patient population:

52 patients will be randomized into two groups in a 2:1 proportion: ph-VEGF-A/FGF (pVIF) treatment group (n=34) and placebo group (n=18). The analysis will be performed on an intention to treat basis.

All patients enrolled in the study will receive optimal medical treatment as judged by treating physician. An effort will be made to modify the medical therapy during the study course only for clear-cut reasons.

Study course and plasmid therapy:

A naked plasmid encoding human or placebo plasmid will be used in the study. The plasmid will be synthesized at the Department of Cell Biology, Cancer Center, Warsaw , Poland by the team of Prof. P. Janik, co-participating in the study. The VEGF-A165 and bFGF cDNA is incorporated into a pSec expression plasmid along with a CMV promoter and zeocin resistance gene and amplified in the E. coli DH5α strain. The plasmid is extracted according to the method described by Y. Isner and approved by the FDA. It has also gained the certificate of the Polish Drugs Institute and acceptance of the Ethical Committee of the Institute of Cardiology for limited clinical trial use.

The plasmid will be given at a total dose of 0.5 mg, 10 injections of 0,2 ml each into the region of reversible ischemia. The process of injecting the solution into each of ten points within the ischemic zone will take 20 to 40 seconds to minimize muscle disruption. This dosage regimen seems efficacious and safe, as documented in the works by Sylvén et al., Laham et al. and Isner et al.

After consenting to take part in the trial, eligible patients will be prepared as for a standard invasive cardiology procedure. Standard angiography and ventriculography will be performed prior to plasmid injection therapy. The ischemic area of interest will be identified on inclusion by SPECT. Cardiac nuclear magnetic resonance (cNMR) with adenosine will also be performed to assess heart morphology, function and perfusion. Next, the injections will be performed according to the protocol described above. The injection catheters supplied by catheter supplied by Johnson&Johnson® (Myo-Star) will be used throughout the study. Proper myocardial needle fixation will be monitored radiographically and on ECG (ventricular extrasystole).

Standard early safety follow-up after injection therapy will include the assessment of basic laboratory parameters (troponin I, CK-MB, RBC, electrolytes), vital signs, echographic evaluation and ECG. Its purpose is to diagnose possible post-injection therapy complications, especially left ventricle puncture or major bleeding.

Follow-up visits will be performed at month 4 and month 12 after injection therapy.

Each visit will include full history, physical examination, laboratory assessment, ECG and exercise test. Dipyridamole-stress SPECT and echocardiographic evaluation will be performed at inclusion and then at month 4 - the time after expected termination of plasmid expression.

At weeks 1, 2, 4, 8 after injection therapy blood samples will be obtained to assess plasma VEGF-A and bFGF levels.

Primarily, a change in myocardial perfusion at rest and on dipyridamole-stress SPECT evaluation after injection therapy will be a measure of efficacy. Changes in exercise tolerance will also be monitored along with a number of other efficacy and safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Severe (>= CCS III) ischemic heart disease despite optimal medical treatment in patients not amenable to percutaneous transluminal coronary angioplasty or coronary artery bypass surgery
* Left ventricular ejection fraction >35%
* Significant stress-induced reversible ischemic area documented on dipyridamole stress myocardial perfusion scintigraphy
* Able to understand and willing to sign the informed consent
* Older than 18 years of age

Exclusion Criteria:

* Angina <CCS III
* Secondary angina
* Acute myocardial infarction within 4 weeks prior to inclusion
* Diabetes with proliferative retinopathy
* Diagnosed or suspected tumor
* Chronic inflammatory or autoimmune disease
* Fertile women
* Left ventricular ejection fraction <35%
* Patients not willing to or not able to give the informed consent to participate in the study
* Patients with a severe disease (other than CAD) having life-expectancy below 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2004-12; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Change in myocardial perfusion at rest and on dipyridamole-stress SPECT evaluation at month 4 after injection therapy | 4 months

SECONDARY OUTCOMES:
Changes in exercise tolerance | month 4 and 12
Changes in life quality and patient's clinical condition | month 4 and 12
Angiographic changes | 4 months
The occurrence of major cardiac adverse events (MACE) during long-term follow-up | throughout the 1-year follow-up
Serum VEGF-A165 and bFGF level | week 1,2,4,8
The occurrence of adverse events related to the plasmid administration procedure | Hospitalization related to procedure
occurrence of adverse events that may be related to overt VEGF or FGF activity | throughout the 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Witold Ruzyllo, Prof., Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, Warsaw, Poland

REFERENCES:
- [Background] Kukula, K., Dabrowski, M., Chojnowska, L., Chmielak, Z., Witkowski, A., Skwarek, M., Kadziela, J., Malecki, M., Teresinska, A., Kownacki, L., Piotrowska-Kownacka, D., Ruzyllo, W., Theoretical base and investigational plan of the VIFCAD study- gene therapy for refractory coronary artery disease in no-option patients using transendocardial bicistronic VEGF/FGF plasmid injection. Post Kardiol Interw; 2, 1 (2006) 116-123
- [Derived] Kukula K, Urbanowicz A, Klopotowski M, Dabrowski M, Pregowski J, Kadziela J, Chmielak Z, Witkowski A, Ruzyllo W. Long-term follow-up and safety assessment of angiogenic gene therapy trial VIF-CAD: Transcatheter intramyocardial administration of a bicistronic plasmid expressing VEGF-A165/bFGF cDNA for the treatment of refractory coronary artery disease. Am Heart J. 2019 Sep;215:78-82. doi: 10.1016/j.ahj.2019.06.009. Epub 2019 Jun 19. PMID 31288177
- [Derived] Kukula K, Chojnowska L, Dabrowski M, Witkowski A, Chmielak Z, Skwarek M, Kadziela J, Teresinska A, Malecki M, Janik P, Lewandowski Z, Klopotowski M, Wnuk J, Ruzyllo W. Intramyocardial plasmid-encoding human vascular endothelial growth factor A165/basic fibroblast growth factor therapy using percutaneous transcatheter approach in patients with refractory coronary artery disease (VIF-CAD). Am Heart J. 2011 Mar;161(3):581-9. doi: 10.1016/j.ahj.2010.11.023. Epub 2011 Jan 31. PMID 21392615